CLINICAL TRIAL: NCT00751491
Title: Randomized Comparison of Adenosin Intracoronary Infusion and Clopidogrel Pretreatment on Myonecrosis Occurence in Elective PCI
Brief Title: Clopidogrel Versus Adenosin in Non Urgent Percutaneous Coronary Intervention (PCI)
Acronym: RACE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: GENNARO SARDELLA, POLICLINICO UMBERTO I-SAPIENZA UNIVERSITY OF ROME
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARD55
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Stable Angina; Percutaneous Coronary Intervention
Keywords: Stable angina; Percutaneous Coronary Intervention; Myonecrosis
MeSH Terms: conditions — Angina, Stable | interventions — Adenosine; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- III (Active Comparator)
  Interventions: Drug: Clopidogrel
- A (Active Comparator)
  Interventions: Drug: Adenosin
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Adenosin — Intracoronary Adenosin 50 microg;
  Other Names: PERCUTANEOUS CORONARY ANGIOGRAPHY
  Arms: A
Other: placebo — no intervention
  Arms: placebo
Drug: Clopidogrel — Clopidogrel 300/600 mg
  Arms: III

SUMMARY:
Percutaneous coronary intervention (PCI) is associated with up to 30% incidence of myonecrosis, as reflected by elevation of cardiac enzymes in a successful procedure. Apart from side-branch occlusion, intimal dissection and coronary spasm, a possible aetiology of myonecrosis after PCI might be distal embolization of atherogenic materials from plaque disruption causing obstruction of blood ﬂow at capillary level resulting in micro-infarction. Recent studies have suggested that pretreatment with adenosine in the cath lab and Clopidogrel and statins greater than 6 hours before may be associated with a reduction in infarct size after reperfusion therapy for acute myocardial infarction. Whether pretreatment with adenosine decreases the incidence of myonecrosis in patients undergoing non-urgent PCI is not fully known. The investigators propose that adenosine-induced hyperaemia can potentially ameliorate the deleterious effects of distal embolization associated with non-urgent PCI through dilatation of the microvasculature. Mechanistically, this may reduce capillary obstruction by facilitating the throughput passage of embolized platelet thrombi out to the venous end of the coronary circulation, thereby reducing the incidence of post-PCI myonecrosis. In this prospective, randomized, open-label study, the investigators evaluated the incidence of myonecrosis after non-urgent PCI with a treatment with intracoronary adenosine compared with pretreatment of loading dose of Clopidogrel 300/600 mg >/< 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Baseline creatine-kinase (CK) and creatine-kinase-myocardial band (CK-MB) had to be within normal limits (a normal CK and CK-MB and elevated troponin allowed inclusion)

Exclusion Criteria:

* Occlusion resulting in Thrombolysis In Myocardial Infarction (TIMI) grade 0 antegrade ﬂow
* Thrombus-laden lesions
* Significant left main coronary stenosis
* Left ventricular ejection fraction 30%
* Inability to give informed consent
* Bradycardia with heart rate below 50 b.p.m.
* Allergy to adenosine
* The occurrence of myo-cardial infarction within one week

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
20% | 12 months

SECONDARY OUTCOMES:
0% | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: GENNARO SARDELLA, MD, Principal Investigator — DEPT.CARDIOLOGY-POLICLINICO UMBERTO I-SAPIENZA UNIVERSITY OF ROME; MASSIMO MANCONE, MD, Study Director — DEPT.CARDIOLOGY-POLICLINICO UMBERTO I-SAPIENZA UNIVERSITY OF ROME
Locations (1):
- Policlinico Umberto I, Rome, Italy